CLINICAL TRIAL: NCT02333045
Title: Characterization and Modulation of Mucosal Immunity for HIV Prevention in Women
Acronym: MIP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Minimal efficacy of maraviroc alone was found in preliminary data analysis of another study.
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Anandi Sheth, Assistant Professor, Emory University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: IRB00074767
Record Dates: First submitted 2015-01-05; First posted 2015-01-07 (Estimated); Results first posted 2017-12-13 (Actual); Last update posted 2018-01-19 (Actual); Status verified 2017-12

CONDITIONS: HIV
Keywords: HIV-negative; Women; At-risk
MeSH Terms: interventions — Emtricitabine, Tenofovir Disoproxil Fumarate Drug Combination; Maraviroc

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Truvada qd (Experimental): Women will be assigned at random Truvada 1 tablet PO daily
  Interventions: Drug: Truvada qd
- Maraviroc 300 qd (Experimental): Women will be assigned at random Maraviroc 300 mg PO daily
  Interventions: Drug: Maraviroc 300 qd

INTERVENTIONS:
Drug: Truvada qd — Truvada 1 tablet PO daily for 7 days
  Other Names: Truvada
  Arms: Truvada qd
Drug: Maraviroc 300 qd — Maraviroc 300 mg PO daily for 7 days
  Other Names: Selzentry
  Arms: Maraviroc 300 qd

SUMMARY:
This study seeks to understand the immune cells in the cervical fluid of in the blood and genital tract of HIV-negative healthy female volunteers and to see if these cells can be modified using a combined anti-viral and antiinflammatory drug called maraviroc, a medicine used in the treatment of HIV infection.

DETAILED DESCRIPTION:
In this study, the investigator seeks to understand the immune cells in the cervical fluid of HIV-negative healthy female volunteers, and to see if these cells can be modified using a combined anti-viral and antiinflammatory drug called maraviroc, a medicine used in the treatment of HIV infection. Maraviroc works by preventing HIV from entering human immune cells by blocking a protein on the outside of these cells called the C-C chemokine receptor type 5 (CCR5) receptor. When maraviroc is bound to this protein, the virus cannot enter the cell. The investigator thinks that CCR5 antagonists could be particularly good drugs for HIV pre-exposure prophylaxis (PrEP) and could potentially be dosed in ways that are easier to take than the current drugs used for PrEP.

In order to further evaluate this PrEP strategy, the investigator will first study the immune cells in the blood and genital tract of HIV-negative healthy female volunteers over the course of 3 months to see how these cells change over time and are affected by factors such as age, menstrual cycle, and genital infections.

The amount of maraviroc compared with the drugs in the current drugs used for PrEP (tenofovir/ emtricitabine) in the blood and genital tract of HIV-negative healthy female volunteers before, during, and after they are given maraviroc versus tenofovir/ emtricitabine for 7 days will be measured. We will also study immune cells from the blood and genital tract from these women to see if maraviroc, tenofovir, or emtricitabine have an effect on these cells that would prevent them from becoming infected with HIV.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-44 years
* Must be biologically female (defined as sex at birth)
* HIV negative women with at least one of the following risk factors in the past 5 years

  1. Injection drug use or use of crack, cocaine, heroin, or methamphetamine
  2. Diagnosed with a sexually transmitted infection
  3. Unprotected sex with 3 or more men
  4. Having sex for drugs, money, or shelter
  5. Sex with a known HIV-positive man
  6. Having a partner meeting any of the preceding criteria
* Normal menses (within 22-35 day intervals) for at least 3 cycles
* No history of alcohol abuse, heart disease, or liver disease, or any other medical condition that would interfere with the conduct of the study, in the opinion of the study investigator
* No history of loop electrosurgical excision procedure (LEEP), conization, or cryosurgery
* Normal chemistry, liver function, and complete blood count panels at screening, including:

  1. Absolute neutrophil count (ANC) ≥ 750/mm3
  2. Hemoglobin ≥ 10.0 g/dL
  3. Platelet count ≥ 100,000/mm3
  4. Aspartate aminotransferase (AST), alanine aminotransferase (ALT), and alkaline phosphatase ≤ 3 x Upper Limit Normal (ULN)
  5. Total bilirubin ≤ 2.5 x ULN
  6. Creatinine Clearance (CrCl) ≥ 60 mL/min as estimated by the Cockcroft-Gault equation
* Negative hepatitis B surface antigen (HBsAg)
* No signs or symptoms of orthostasis
* No signs or symptoms of vaginal infection or genital ulcer disease at screening or untreated vaginal infection in the last 30 days
* Not receiving concurrent medications that interact with maraviroc (MVC) or any antiretrovirals (such as tenofovir/ emtricitabine [Truvada®]) for the purpose of HIV prevention
* Willing to use condoms for the duration of the study and abstain from sexual intercourse for 48 hours before each genital tract sampling

Exclusion Criteria:

* Male sex (defined as sex at birth)
* Pregnant or breastfeeding
* Current use of systemic hormonal contraception
* Symptomatic vaginal infection or genital ulcer disease at screening or treatment for vaginal infection in the last two weeks
* Active malignancy for which the participant is undergoing evaluation and/or treatment
* Immunosuppressive medications (i.e, systemic steroids)
* Any surgery in the preceding 2 months

Ages: 18 Years to 44 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 4 (Actual)
Dates: Start 2015-01; Primary Completion 2016-10-28 (Actual); Study Completion 2016-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anandi Sheth, MD, Principal Investigator — Emory University
Locations (2):
- United States (2):
  - Grady Memorial Hospital, Atlanta, Georgia
  - Grady Infectious Diseases Clinic (Ponce Clinic), Atlanta, Georgia

RESULTS

PARTICIPANT FLOW:
Groups:
- Truvada: Women randomized to receive one tablet of Truvada (200mg emtricitabine/300mg tenofovir) daily for 7 days.
- Maraviroc: Women randomized to receive 300mg of Maraviroc daily for 7 days.
Period: Overall Study
Arm/Group | Truvada | Maraviroc
Started | 1 | 3
Completed | 1 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: All individuals who gave informed consent to participate in the study and who met eligibility criteria are included in the baseline analysis description.
Groups:
- Total: Total of all reporting groups
Arm/Group | Truvada | Maraviroc | Total
Number analyzed (Participants) | 1 | 3 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 3 | 4
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 1 | 3 | 4
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 3 | 3
  White | 1 | 0 | 1
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1 | 3 | 4

OUTCOME MEASURES:

1. Primary Outcome: Count of Total Cells Obtained From Cervicovaginal Lavage Samples
Description: The count of CCR5+CD4+ T cells in the genital tract, before participants began study treatment, after 7 days of treatment, and during the post-treatment drug elimination period. The precise role of CCR5+CD4+ T cells in the female genital tract is unknown, however, higher cell counts may suggest the potential for more HIV target cells in the genital tract.
Time Frame: Baseline, Day 7, Day 14, Day 21
Population: The analysis includes all available data collected during each study visit. Not all participants provided a sample at every study visit.
Measure: Mean (Standard Deviation); unit: cells
Arm/Group | Truvada | Maraviroc
Number analyzed (Participants) | 1 | 3
cells
  Baseline: number analyzed (Participants) | 1 | 1
  Baseline | 42,000,000 (0.0) | 20,000,000 (0.0)
  Day 7: number analyzed (Participants) | 1 | 2
  Day 7 | 15,000,000 (0.0) | 18,700,000 (7,500,000)
  Day 14 | 20,000,000 (0.0) | 28,300,000 (8,500,000)
  Day 21 | 30,000,000 (0.0) | 21,800,000 (13,200,000)

2. Secondary Outcome: Steady-state Area Under the Plasma Concentration-time Curve of Study Drug
Description: Study drug concentrations will be measured from blood.
Time Frame: 7 days
Population: Data were not collected at each visit as some participants declined providing samples. Due to the small number of observations, study drug concentrations were not determined for the samples provided.
Arm/Group | Truvada | Maraviroc
Number analyzed (Participants) | 0 | 0

3. Secondary Outcome: Steady-state Area Under the Female Genital Tract Concentration-time Curve of Study Drug
Description: Study drug concentrations will be measured from female genital tract.
Time Frame: 7 days
Population: as for outcome 2
Arm/Group | Truvada | Maraviroc
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Adverse events were recorded during the entire duration of participation for each individual subject, from signing the consent form through the 21 day follow up period.
Description: Genitourinary symptoms will be recorded at each visit. Signs and symptoms will be graded according to the Division of AIDS Table for Grading the Severity of Adult and Pediatric Adverse Events (DAIDS AE Grading Table), Version 1.0, December 2004.
Groups:
- Truvada: Women randomized to receive on tablet of Truvada daily for 7 days.
- Maraviroc: Women randomized to receive 300mg of Maraviroc 300 mg daily for 7 days.
Arm/Group | Truvada | Maraviroc
All-Cause Mortality (participants affected / at risk) | 0/1 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/1 | 0/3
Other Adverse Events (participants affected / at risk) | 0/1 | 0/3

LIMITATIONS AND CAVEATS:
In 2016, preliminary data analyses of a prior study and similar trials suggested minimal effects of a standard dose of maraviroc alone on cells of the female genital tract. Thus this intervention was discontinued early to minimize participant burden.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes